CLINICAL TRIAL: NCT02072135
Title: Exparel Use for Popliteal Nerve Block in Postoperative Pain Control; After Ankle Fracture Fixation or Ankle Fusion Surgery: a Case Series
Brief Title: Exparel and Ankle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013003841
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Ankle Fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exparel (Experimental): Exparel 266mg
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel
  Other Names: liposomal bupivacaine

SUMMARY:
This study involves a drug called Exparel that has been approved by the US Food and Drug Administration (FDA), for application directly to wound sites. EXPAREL® is a long acting pain reliever. It is being given in this study to see if it provides safe and effective pain relief after ankle surgery. Because it is a long acting drug, it may lessen pain relief for as much as 72 hours after surgery.

EXPAREL® has not been approved by the FDA for administration by popliteal block, which is the method the study doctors will use to give the patients the drug. Giving the drug by popliteal block involves inserting a small tube in to the back of the knee to deliver the drug. The study doctors wish to determine if patients undergoing ankle surgery and receiving this drug have less pain and less need for narcotic medication.

DETAILED DESCRIPTION:
Managing postoperative pain remains a paramount topic in anesthesiology, since a significant amount of patients continue to report discomfort after their inpatient and outpatient surgeries. Orthopedic lower limb surgeries are known to induce prolonged pain after the procedure requiring the increased use of multi-modal analgesia. Popliteal fossa nerve block targeting the sciatic nerve has been utilized to effectively control postoperative pain and to lower opioid requirements for patients undergoing foot and ankle surgeries.The sciatic nerve divides into its tibial and common fibula branches approximately 4 to 13 centimeters above the popliteal crease. The tibial nerve innervates the heel and the plantar aspect of the foot, while the common fibula nerve, also known as the common peroneal nerve, supplies the lateral aspect of the leg and the dorsum of the foot.

Bupivacaine, a local anesthetic and analgesic, is currently used as an agent to address postsurgical analgesia. However, administering a large dose of bupivacaine for nerve blockade has been reported to lead to complications such as infection, hematoma, vascular puncture, toxicity and, even severe systemic side effects. EXPAREL® (multi-vesicular liposomal bupivacaine) is a multi-vesicular liposomal form (DepoFoam drug delivery systems) of encapsulated bupivacaine that allows for the slow diffusion of the drug over an extended period of time of 72 hours, versus the 8 hour duration of Bupivacaine Hydrogen Chloride (HCl). EXPAREL® has been shown to provide successful prolonged analgesia after wound infiltration during several surgical procedures.In addition to the long lasting pain relief, studies also highlight the improved clinical outcomes of patients and lower economic costs associated with liposomal bupivacaine when compared to bupivacaine Hydrogen chloride. However, studies evaluating the use of EXPAREL® for nerve blocks are limited. Richard et. al. demonstrated the safety of EXPAREL® to Bupivacaine and saline on the brachial plexus of dogs and rabbits revealing no irritation or tissue damage even at high doses. Furthermore, after administering liposomal bupivacaine via single epidural injections into humans, Viscussi et. al. reported longer sensory blockade and shorter motor blockade compared to bupivacaine HCl, enabling quicker recovery and mobility for the patient.

The primary objectives of this study is to (1) evaluate the efficacy of the study drug EXPAREL® with respect to the safety and duration of the postoperative analgesic effect on five subjects following single dose injection via a popliteal nerve block. Based on the data analysis from this case series, a decision will be made as to whether a large randomized, double-blinded, prospective study is warranted.

Methods and Materials The purpose of the popliteal nerve block with the use of EXPAREL® will be explained to the potential subject. Demographic information will be obtained including age, gender, past medical history, past surgical history, hospitalizations, current medications, allergies, and history of drug and alcohol abuse. Preoperative baseline pain score, motor strength and sensation will be documented by a study team member, prior to carrying out study procedures. The Visual Acuity Scale (VAS) will be explained to the patient. A Semmes Weinstein monofilament exam with a size 5.07 monofilament will be performed to rule out any occult nerve injury.

On the day of surgery all eligible subjects will receive a single dose of study drug EXPAREL® 1.3% 20 ml (266mg) will be administered within 1 hour prior to the surgical procedure as a popliteal nerve block. This block will be done by a trained anesthesiologist, using an ultrasound-guided technique (Mindray model # M-7). Prior to induction of anesthesia, standard monitoring devices such as non-invasive blood pressure, EKG and pulse oximetry for oxygen saturation will be started. Bispectral Index (BIS) will be maintained in a range of 30-60. Continuous vital sign monitoring will be done intraoperatively. All patients will be administered midazolam 0.5 mg to 4 mg/kg to achieve anxiolysis. Induction of anesthesia will also include Lidocaine 1.5mg/kg, Propofol 1.5-3 mg/kg, Fentanyl 1-2mcg/kg. If indicated the muscle relaxant of the anesthesiologists choice: either Succinylcholine 1.5 mg/kg, Rocuronium 0.6mg/kg or Nimbex 0.2mg/kg to titrate Train of Four (TOF) at 1-2 twitches until 30 minutes prior to the end of the surgical procedure. Anesthestic maintenance with 0.8 to 1.5 Minimum Alveolar Concentration (MAC) of sevoflurane as indicated by end tidal concentration in oxygen and air mixture of 50% each and fraction of inspired oxygen ( FiO2) may be increased if oxygen saturation is less than 96%. The use of fentanyl will be permitted during surgery. However, intraoperative administration of any other narcotics or analgesics (including intrathecal opioids), local anesthetics, or anti-inflammatory agents is prohibited, unless needed to treat an adverse even (AE). The amount of fentanyl used will be recorded. Ondansetron0.1mg/kg will be used as an antiemetic prior to reversal of muscle relaxant with neostigmine and glycopyrrolate.

Upon extubation, the patient will be transferred to the post-anesthesia care unit (PACU). At this time quality of the regional block will be assessed. Motor strength will be rated as follows: 2=no voluntary movement, 1=some muscle weakness and 0=no muscle weakness. The sensory block (cold test) will be evaluated by the following criteria: 2=no sensation, 1=decreased sensation and 0=normal sensation. All blocks rated as 0 for both sensory and motor testing, will be considered failed blocks and will be excluded from the data collection for the remainder of the study.

All subjects will receive rescue medication upon request for pain control whether they remain in the data collection or not. Patients will be treated with intravenous Hydromorphone 0.5mg for a pain score ≥ 4 out of 10 on the VAS scale for a maximum of 2 divided doses. Vital signs (heart rate, blood pressure, respiratory rate and pulse oxymetry) will be continuously monitored in the Post Anesthesia Care Unit (PACU) and recorded as to the standard protocol that is every 5 minutes for the first 15 minutes, 15 minute intervals for the next hour and then every 30 minutes until discharge. Pain score and sedation scores will be obtained using the VAS and Ramsay sedation scale, respectively. All pain scores will be assessed with patient in the resting position. No patient will be discharged from the PACU with a VAS >than 4 out of 10. If this cannot be achieved with the rescue medication indicated above the patient will be started on Patient Controlled Analgesia (PCA). PCA orders are as follows Hydromorphone 0.02mg every 6 minutes, no basal rate, and no four-hour maximum. Neurological and sensory assessment will be assessed on arrival, at 60 minutes and at 120 minutes. Those parameters assessed will include numbness of tongue, lips and mouth, metallic taste, problems with hearing or vision, muscle twitching and does the subject feel cold in the innervated dermatomes.

Time to discharge readiness from PACU will be documented. After PACU discharge oxycodone 5mg/325mg acetaminophen 1 or 2 tablets every 6 hours will be offered for breakthrough pain. The doses and timing of all pain medications will be recorded while hospitalized and the subject's will be provided a diary to record pain and medication taken at home. The research coordinator will follow-up with the patients on post-operative days for those who have been discharged to home, in order to ensure that questionnaires and diaries are completed.

On POD 1, POD 2 and POD 3, a pain questionnaire will be completed addressing the quality of postoperative pain relief, pain scale, and incidence and severity of any side effects, including palpitations, nausea, vomiting as well as burning, numbness, tingling, and rebound pain. Peripheral neuropathy sequelae will be assessed subjectively via the questionnaire. The subject will also be evaluated for amount of pain medication required and any opioid side effects will be documented. On POD 3 the subject will be asked to provide an overall opinion of the pain control using a 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* ankle fracture open reduction or internal fixation
* American Society of Anesthesiologists rating of I-III
* have a working telephone

Exclusion Criteria:

* non English speaking
* BMI >40
* allergy or contraindication to local anesthetics
* history of drug abuse
* impaired kidney function, rheumatoid arthritis or loss of sensation in extremities
* abnormal liver function
* long term (greater than 10 days) use of NSAIDS
* uncontrolled anxiety, psychiatric or neurological disorder that might interfere with study assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
pain | 72 hours post operation
  Subject will be asked highest pain score and amount of narcotics used

SECONDARY OUTCOMES:
side effect of drug | 72 hours
  -numbness of lips, tongue or mouth metallic taste in the mouth muscle twitching problems with vision or hearing

CONTACTS AND LOCATIONS:
Overall Officials: Jean Daniel Eloy, MD, Principal Investigator — Rutgers University
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No